CLINICAL TRIAL: NCT00989625
Title: An Open Label, Single Dose, Randomised, Parallel Group Pharmacokinetic Study to Evaluate a Combination Product Containing Naproxen Sodium and Sumatriptan in Adolescent Subjects With Migraine and Healthy Adult Subjects Administered at Three Doses.
Brief Title: A Pharmacokinetic Study to Evaluate TREXIMET in Adolescents With Migraine and Healthy Subjects Administered at Three Doses.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 108504
Record Dates: First submitted 2009-03-20; First posted 2009-10-05 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Migraine Disorders
Keywords: migraine; single dose; healthy volunteer; adolescence; pharmacokinetics
MeSH Terms: conditions — Migraine Disorders | interventions — sumatriptan-naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 10mg Sumatriptan/60mg Naproxen (Active Comparator): There is only one dose (one tablet) for each subject. Subject to be randomized to either: 10mg Sumatriptan/60 mg Naproxen or 30mg Sumatriptan/180mg Naproxen or 85mg Sumatriptan/500mg Naproxen.
  Interventions: Drug: This is a pharmacokinetic study (Treximet)
- 30mg Sumatriptan/180mg Naproxen (Active Comparator): There is only one dose (one tablet) for each subject. Subject to be randomized to either: 10mg Sumatriptan/60 mg Naproxen or 30mg Sumatriptan/180mg Naproxen or 85mg Sumatriptan/500mg Naproxen.
  Interventions: Drug: This is a pharmacokinetic study (Treximet)
- 85mg Sumatriptan/500mg Naproxen (Active Comparator): There is only one dose (one tablet) for each subject. Subject to be randomized to either: 10mg Sumatriptan/60 mg Naproxen or 30mg Sumatriptan/180mg Naproxen or 85mg Sumatriptan/500mg Naproxen.
  Interventions: Drug: This is a pharmacokinetic study (Treximet)

INTERVENTIONS:
Drug: This is a pharmacokinetic study (Treximet) — This is a pharmacokinetic study to collect PK samples from subject after single dose.
  Arms: 10mg Sumatriptan/60mg Naproxen
Drug: This is a pharmacokinetic study (Treximet) — This is a pharmacokinetic study to collect PK samples from subject after single dose.
  Arms: 30mg Sumatriptan/180mg Naproxen
Drug: This is a pharmacokinetic study (Treximet) — This is a pharmacokinetic study to collect PK samples from subject after single dose.
  Arms: 85mg Sumatriptan/500mg Naproxen

SUMMARY:
This is a pharmacokinetic (PK) study designed to investigate a combination product containing sumatriptan succinate and naproxen sodium administered at 3 single doses (10mg sumatriptan/60mg naproxen sodium, 30mg sumatriptan/180mg naproxen sodium, 85mg sumatriptan/500mg naproxen sodium) in adolescent migraine patients. The same doses will be also administered to a group of healthy volunteer (HV) adult subjects and the PK parameters will be compared between these two groups and between doses.

DETAILED DESCRIPTION:
This will be an open label, single dose, randomised, parallel group study. Approximately 27 adolescent patients with migraine and 27 healthy volunteer (HV) adult subjects will be enrolled so that a total of 24 evaluable subjects complete in each group. The treatment procedures for these two groups are almost identical but some flexibility has been allowed for the timing of some of the PK samples in adolescents. All subjects will be required to attend a screening visit within 28 days prior to the first dose of study medication. Each subject will participate in one dosing session with one of the 3 doses of sumatriptan/ naproxen sodium. Sequential PK samples will be collected through 48 hours after dosing and the PK parameters will be compared between these two groups and between doses.

ELIGIBILITY:
Inclusion Criteria:

Adolescent Migraine Subjects

* Subject has history of migraine with or without aura.
* Subject has history suggestive of typical migraine attacks with duration of about 2 or more hours.
* Subject has at least 2, but not more than 8, migraine attacks per month in each of the 2 months prior to the screening visit.
* Subject has at least a 6-month history of moderate to severe migraine attacks, sufficient to establish a definitive diagnosis of migraine.
* Subject is able to distinguish migraine from other headaches (e.g., tension-type headaches).

All subjects

* Subject must fall between following age ranges:

  * Adolescent subjects between 12 and 17 years old inclusive at the screening visit and 18 years at dosing.
  * Adult healthy subjects between 18 to 55 years old inclusive at the screening visit.
* Subject BMI and weight must fall between the following:

  * Adolescent subject body weight less than 33.4 kg and a healthy weight using age-based BMI range 5th-85th percentile (see Appendix 4).
  * Adult healthy subject BMI within the range 18-32 kg/m2 inclusive
* Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and ECG. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* A female subject is eligible to participate if she is of:

  * Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory]. For younger adolescent migraine subjects, non-childbearing potential also defined as premenarchal is a young female who has not yet entered puberty as evidenced by lack of breast development of palpable glandular breast tissue. Females on hormone replacement therapy and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1 if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.]
  * Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects who are sexually active must agree to use contraception until 5 day after dosing.
* Subjects must be able to read and write English or Spanish and give written informed consent as follows:

  * Adult: subject is willing and able to provide written informed consent
  * Adolescent: subject is capable of giving written assent with an informed consent from their parents or legal guardian, which includes compliance with the requirements and restrictions listed in the consent form.
* Eligible subjects should meet the QT criteria as follows:

  * Adolescent: QTcB or QTcF <450 msec; and without Bundle Branch Block
  * Adult: QTcB or QTcF<450 msec; or QTc <480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

Adolescent Migraineur Subjects

* Subject has ≥15 headache days per month in total, retinal, basilar or hemiplegic migraine or secondary headaches.
* Subject is experiencing a migraine attack or has experienced a migraine attack within 24 hours of dosing.

All subjects:

* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive test for HIV antibody.
* Subject, in the investigator's opinion, is likely to have unrecognized cardiovascular or cerebrovascular disease (See Appendix 1)
* Subject has uncontrolled hypertension

  * Adults: systolic >/=140 mmHg, diastolic >/=90mmHg
  * Adolescent BP >/= 95 percentile adjusted for age, height and gender (Appendix 4).
* Subject has a history of congenital heart disease, cardiac arrhythmias requiring medication, or a history of a clinically significant electrocardiogram abnormality that, in the investigator's opinion, contraindicates participation in this study.
* Subject has evidence or history of any ischemic vascular diseases including:ischemic heart disease, ischemic abdominal syndromes, peripheral vascular disease or Raynaud's Syndrome, or signs/symptoms consistent with any of the above.
* Subject has evidence or history of central nervous system pathology including stroke and/or transient ischemic attacks, epilepsy or structural brain lesions which lower the convulsive threshold; or has been treated with an antiepileptic drug for seizure control within 5 years prior to screening.
* Subject has a history of impaired hepatic or renal function
* Subject has hypersensitivity, allergy, intolerance, or contraindication to the use of any triptan, NSAID or aspirin (including all sumatriptan and naproxen preparations) or has nasal polyps and asthma.
* Subject is currently taking, or has taken in the previous three months, a migraine prophylactic medication containing methysergide or dihydroergotamine; or is taking a medication that is not stabilized (i.e., change of dose within the past month) for either chronic or intermittent migraine prophylaxis or for a co-morbid condition that is not stabilized.
* Subject has a recent history of regular use of opioids or barbiturates for treatment of his/her migraine headache and/or other non-migraine pain. Regular use is defined as an average of 4 days per month over the last 6 months.
* Subject has taken, or plans to take, a monoamine oxidase inhibitor, or herbal preparations containing St. John's Wort (Hypericum perforatum), anytime within the 2 weeks prior to screening through 2 weeks post final study treatment.
* Subject history of any bleeding disorder or is currently taking any anti-coagulant or any anti-platelet agent.
* Subject has evidence or history of any gastrointestinal surgery (other than appendectomy >/=6 months previously which is permitted) or GI ulceration or perforation or gastrointestinal bleeding or evidence or history of inflammatory bowel disease.
* Subject is pregnant, actively trying to become pregnant, or breast feeding or subject not willing to have pregnancy test performed at each study visit.
* Sexually active female subjects using inadequate contraceptive measures (i.e., a method with a failure rate >1%)
* Subject has evidence of alcohol or substance abuse within the last year or any concurrent medical or psychiatric condition which, in the investigator's judgment, will likely interfere with the study conduct, subject cooperation, or evaluation and interpretation of the study results, or which otherwise contraindicates participation in this clinical trial.
* History of regular alcohol consumption within 6 months of the study defined as:

  * Adults: An average weekly intake of >14 drinks/week for men or >7 drinks/week for women. One drink is equivalent to (12 g alcohol) = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits.
  * Adolescents: Adult limits may be applicable for adolescents >16 years of age. For adolescents in younger group (< 16 years of age) that enrolment will be at the discretion of the investigator, but drinking should be no more than 50% of the allowance for adults (e.g. children of 14 are drinking no more than 7 drinks (70 g week, [Tur, 2003]).
* Subject has participated in an investigational drug trial within the previous 4 weeks or plans to participate in another study at any time during this study.
* An adult subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer). An adolescent subject should not have received an investigational product within the previous 6 months.
* Subject exposure to chemical entities defined as:

  * Adult subject exposed to more than four new chemical entity within 12 months prior to the first dosing day.
  * Adolescent subject exposed to more than 1 new chemical entities within 12 months prior to the first dosing day
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Subjects would have made a total donation of blood or blood products in excess of the following:

  * 500 mL within a 56 day period before screening for Healthy adult subjects
  * 10mL/kg within a 56 day period before screening for adolescents
* Unwillingness or inability to follow the procedures outlined in the protocol
* Subjects who are kept due to regulatory or juridical order in an institution.

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2008-11-04 (Actual); Primary Completion 2009-09-10 (Actual); Study Completion 2009-09-10 (Actual)

PRIMARY OUTCOMES:
To compare the pharmacokinetics of naproxen sodium and sumatriptan following the administration of the combination tablet at 3 doses (10mg sumatriptan/60mg naproxen, 30mg sumatriptan/180mg naproxen, 85mg sumatriptan/500mg naproxen) from 0 to 48 hours. | Derived pharmacokinetic parameters including AUC(0-2), AUC(0-Inf), AUC(0-t) and Cmax for sumatriptan at each dose. Derived pharmacokinetic parameters including AUC(0-Inf), AUC(0-t) and Cmax, for naproxen at each dose from 0 to 48 hours.

SECONDARY OUTCOMES:
To investigate the safety and tolerability of the combination tablet at 3 doses in adolescent migraine subjects and healthy adult subjects over 2 weeks. | Derived PK parameters including tmax, t½, and Cl/F (0-48 hours) for sumatriptan at each dose. Derived pharmacokinetic parameters including tmax and t½ and Cl/F for naproxen sodium at each dose. Reported AEs, BP, heart rate, 12-Lead (0-48 hours).
Report adverse events, blood pressure, heart rate and 12-Lead ECG over 2 weeks. | These will be measured after dosing within 48 hours and 7-14 days after dosing period.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 108504 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/108504?search=study&study_ids=108504#rs
- Available data/document: Study Protocol: 108504 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 108504 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 108504 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 108504 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 108504 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 108504 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 108504 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register